CLINICAL TRIAL: NCT04890613
Title: Phase Ib Expansion Study of CX-5461 in Patients With Solid Tumours and BRCA2 and/or PALB2 Mutation
Brief Title: Study of CX-5461 in Patients With Solid Tumours and BRCA1/2, PALB2 or Homologous Recombination Deficiency (HRD) Mutation
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Senhwa Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CX-5461-04
Record Dates: First submitted 2021-05-05; First posted 2021-05-18 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Tumor
Keywords: Pancreatic Cancer; Ovarian Cancer; Prostate Cancer; Breast Cancer; BRCA1 and/or other HRD-associated mutation; somatic or germline BRCA1/2 and/or PALB2 mutation
MeSH Terms: conditions — Pancreatic Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms; Breast Neoplasms | interventions — CX 5461

STUDY DESIGN:
Intervention Model Description: Eligible patients will be enrolled into two cohorts; Main study cohort: Patients with histologically-confirmed pancreatic, ovarian, prostate, or breast cancers with pathogenic/likely pathogenic germline or somatic BRCA1/2, PALB2, and/or other specified genetic alterations. Exploratory cohort: women with ovarian cancer and pathogenic/likely pathogenic BRCA1 and/or other HRD-associated mutation.
  An initial 16 eligible patients for the main cohort and 10 eligible patients for the exploratory cohort will be enrolled to receive CX-5461 at 250mg/m2, delivered as a 60-minute IV infusion on Day 1 and Day 8 of a 28-day cycle. Upon completion of enrollment of all patients in the initial arms, if there are no safety concerns after review of the safety data, another two arms will open to enroll an additional 16 patients for the main cohort and 10 patients for the exploratory cohort to receive CX-5461 at 325mg/m2, delivered as a 60-minute IV infusion on Day 1 and Day 8 of a 28-day cycle.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Main Study Cohort patients receiving CX-5461 at 250mg/m2 (Experimental): Eligible patients with histologically confirmed pancreatic, ovarian, prostate, or breast cancers with pathogenic/likely pathogenic germline or somatic BRCA1/2 and/or PALB2 mutation and/or genetic alterations in the specified genes will be enrolled to receive CX-5461 at a dosing concentration of 250mg/m2, delivered as a 60-minute IV infusion on Day 1 and Day 8 of a 28-day cycle.
  Interventions: Drug: CX-5461
- Exploratory cohort patients receiving CX-5461 at 250mg/m2 (Experimental): Eligible patients with ovarian cancer and pathogenic/likely pathogenic BRCA1 and/or other HRD-associated mutation will be enrolled to receive CX-5461 at a dosing concentration of 250 mg/m2, delivered as a 60-minute IV infusion on Day 1 and Day 8 of a 28-day cycle.
  Interventions: Drug: CX-5461
- Main Study Cohort patients receiving CX-5461 at 325mg/m2 (Experimental): After confirming the dose of 250mg/m2 to be safe and tolerable, eligible patients with histologically confirmed pancreatic, ovarian, prostate, or breast cancers with pathogenic/likely pathogenic germline or somatic BRCA1/2 and/or PALB2 mutation and/or genetic alterations in the specified genes will be enrolled to receive CX-5461 at a dosing concentration of 325mg/m2, delivered as a 60-minute IV infusion on Day 1 and Day 8 of a 28-day cycle.
  Interventions: Drug: CX-5461
- Exploratory cohort patients receiving CX-5461 at 325mg/m2 (Experimental): After confirming the dose of 250mg/m2 to be safe and tolerable, eligible patients with ovarian cancer and pathogenic/likely pathogenic BRCA1 and/or other HRD-associated mutation will be enrolled to receive CX-5461 at a dosing concentration of 325 mg/m2, delivered as a 60-minute IV infusion on Day 1 and Day 8 of a 28-day cycle.
  Interventions: Drug: CX-5461

INTERVENTIONS:
Drug: CX-5461 — 150 mg sterile lyophilized powder containing 1% sucrose
  Other Names: Pidnarulex

SUMMARY:
This is an open-label, multi-center, phase 1b study designed to determine a tolerable dose of CX-5461 administered by IV infusion on Day 1 and Day 8 of a 28-day cycle in patients with selected solid tumours and associated mutations for future Phase II trials. The safety and tolerability of CX-5461, preliminary evidence of antitumor effect and the effect of CX-5461 on the Health-Related Quality of Life (HRQoL) will also be evaluated. The study will also evaluate the predictive value of mutational signatures and explore the significance of dynamic changes in ctDNA levels and plasma DNA methylome profiling in this study's exploratory cohort.

DETAILED DESCRIPTION:
CX-5461 (Pidnarulex), a synthetically-derived small molecule that selectively kills HR-deficient cancer cells through the binding and stabilization of G4 DNA structure. Early phase 1 studies suggest CX-5461 has activity and warrants further investigation in HR-deficient tumors. This study aims to determine the tolerable dose of CX-5461 for phase II studies, amongst an expansion cohorts of BRCA1/2, PALB2 or HRD mutant tumors.

ELIGIBILITY:
Inclusion Criteria:

Main study cohort:

1. Histologically or cytologically confirmed malignancy of the pancreas, prostate, breast, or ovary.
2. Documented evidence of pathogenic or likely pathogenic somatic or germline mutation in BRCA1/2 and/or PALB2, and/or any genetic alterations listed below as indicated in a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory report. The report must be submitted to and approved by study sponsor prior to registration. Other HRD-associated mutations could be eligible if prior approval by the sponsor is granted.

ATM, ATR, BARD1, BRCA1, BRCA2, BRIP1, CCNE1, CHEK1, CHEK2, CDK12, CREBBP, FANCA, FANCI, FANCL, FANC2, FANCB, FANCC, FANCD2, FANC family*, MRE11A, MYC, NBN, NCL, PALB2, RAD50, RAD51B, RAD51C, RAD51D, RAD54L, SLFN11, PTIP, MLL3, MLL4, EZH2, CtIP(RBBP8), MUS81, CDH4, DYNLL11, TOPBP1, NBS1, CDC25A, CDC25C, RAD17, WEE1

* In addition to the genes already specified, the "FANC family" genes may also include the following: FANCE, FANCF, FANCG, FANCM, FANCP, FANCQ/ERCC4/XPF, FANCR/RAD51, FANCT/UBE2T, FANCU/XRCC2, FANCV/REV7/MAD2L2, and FANCW/RFWD3.

Exploratory cohort:

1. Histologically confirmed ovarian, fallopian tube or primary peritoneal cancer, with a high grade serous or high grade endometrioid histology subtype.
2. Documented evidence of pathogenic or likely pathogenic germline mutation or a clinically actionable somatic mutation in BRCA1 and/or other HRD-associated mutation, as indicated in a CLIA-certified laboratory report. The report must be submitted to and approved by study sponsor prior to registration.
3. Meet one of the following criteria:

   1. Platinum Sensitive with no evidence of disease progression within 6 months of the last dose of platinum-based chemotherapy (n=10 patients); OR
   2. Platinum Resistant with disease progression within 6 months of the last dose of a platinum-based chemotherapy.

All participants:

1. Age ≥ 18 years.
2. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 within 14 days of registration.
3. Radiographically documented disease progression within 28 days of registration and evaluable as per RECIST v1.1.
4. Patient must have measurable disease as per RECIST v1.1.
5. Patients must have adequate bone marrow, renal and hepatic function per local laboratory reference ranges as follows within 14 days of registration:

   1. Absolute Neutrophil Count ≥ 1.5 x 10^9/L
   2. Platelets ≥ 100 x 10^9/L
   3. Hemoglobin ≥ 9 g/dL (blood transfusion ≤ 7 days of screening not permitted).
   4. Calculated creatinine clearance > 51mL/min (Cockcroft-Gault formula)
   5. AST/ALT ≤ 2.5× the upper limit of normal (ULN). Subjects with liver metastasis may have AST, ALP, and ALT ≤ 5.0 X ULN.
   6. Bilirubin ≤ 1.5×ULN. This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of haemolysis or hepatic pathology), who will be allowed only at the discretion of the Study Investigator.
   7. INR/PT and aPTT ≤1.5 X ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
   8. Albumin ≥3.0 g/dL
6. Patients are willing to undergo tumour biopsy pre-treatment and at time of progression on treatment. If a biopsy at the time of progression on prior therapy is available and can be submitted to the Central Lab for this study, this procedure does not need to be repeated. Patients who consent but have tumour that is not amenable to safe biopsy will be allowed to enter the trial and continue therapy as per protocol if this has been addressed and permission is granted from the sponsor prior to registration.
7. Life expectancy of greater than 3 months from the date of registration.
8. Able to provide written informed consent.
9. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
10. Female patients of childbearing potential must have a negative serum pregnancy test within 14 days prior to registration. (Note: a negative urine/serum pregnancy test is required on Cycle 1, Day 1 prior to treatment unless the screening pregnancy test was done within 48hrs of registration).
11. Female patients of childbearing potential and male patients who are sexually active must agree to practice true abstinence or at least two effective methods of contraception (ie: condoms with spermicide, hormonal methods such as oral contraceptive pills, vaginal ring, injectables, implants and intrauterine devices (IUDs), non-hormonal IUDs, such as ParaGard, bilateral tubal ligation, vasectomy, complete abstinence) within 14 days prior to registration, and agree to continue using such precautions while on treatment with CX-5461 (including dose interruptions) and for 6 months following the last dose of CX-5461.
12. There is no minimum or maximum number of lines of prior therapy and prior PARP inhibitor therapy is allowed.
13. Patient is clinically stable at the time of entering the study.

Exclusion Criteria:

1. For pancreatic cancer; non-adenocarcinoma histology is excluded from this study.
2. Patients with malignant bowel obstruction.
3. Untreated, unstable brain or meningeal metastases or tumor. Patients with radiological evidence of stable brain metastases are eligible provided that they are asymptomatic and either do not require corticosteroids or have been treated with corticosteroids, with clinical and radiological evidence of stabilization at least 10 days after discontinuation of steroids.
4. Unresolved toxicity > CTCAE grade 1 from previous anti-cancer therapy (including radiotherapy) except hematological toxicity, Grade 1 or 2 neuropathy, and alopecia.
5. Any evidence of severe or uncontrolled diseases such as but not limited to active infection, unstable or uncompensated respiratory, cardiac, neurological, hepatic, renal disease or psychiatric illness/social situations, which in the opinion of the investigator, would limit compliance with study requirements.
6. Treatment with an investigational (non-registered - other than PARP inhibitor) agent within 30 days and treatment with PARP inhibitor within 14 days prior to the first dose of study medication.
7. Immuno-compromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV), patients with known active hepatitis (i.e., hepatitis B or C). Note: Patients with a prior history of treated HBV infection who are antigen-negative or patients with a prior history of treated HCV infection who are HCV RNA-undetectable may be enrolled. Patients who are known to be serologically positive for human immunodeficiency virus (HIV) can enroll if their CD4+ T-cell (CD4+) counts ≥ 350 cells/uL.
8. Patients who have had recent (within 14 days of registration, or until any wound has completely healed) major thoracic or abdominal surgery prior to study start, or a surgical incision that is not fully healed.
9. No concurrent systemic anti-cancer therapy, biological therapy or other novel agent is to be permitted. Palliative radiotherapy may be allowed. If radiotherapy is required due to disease progression, patient will be considered off study. If radiotherapy is be used to treat non-target lesions and patients may benefit from continuing on study treatment, CX-5461 may re-commence 14 days after completion of radiotherapy. Any continuation on study treatment must be discussed with and approved by study sponsor.
10. Patients may be potentially eligible where the current tissue diagnosis is confirmed histologically from biopsy of a target lesion, and the patient has had no evidence of active second malignancy which requires treatment or would confound interpretation of safety, tolerability and efficacy of CX-5461. These cases must be discussed with the medical monitor prior to confirm eligibility.
11. Presence of known photosensitivity disorders (xeroderma pigmentosa, porphyria etc.). Strict adherence to protocol-defined sun-protection measures is essential for the duration of study. Patients who do not agree to follow these measures are not eligible. Patients who do not agree to use sunglasses and sun blocker (with SPF50 to UVB and a high degree of protection against UVA) if exposed to sunlight during the course of the study and for 3 months after the last dose are not eligible. Patients who plan to use sunbeds or tanning booths during the course of the study and within 3 months after the last dose are not eligible.
12. Female patients who are pregnant or nursing.
13. Ophthalmological active ocular surface disease at baseline (based on ophthalmological evaluation).
14. History of cicatricial conjunctivitis (as evaluation by an ophthalmologist).
15. Has had radiotherapy with a limited field for palliation within 1 week of the first dose of study drug, with the exception of patients receiving radiation to more than 30% of the bone marrow or with a wide field of radiation, which must be completed at least 4 weeks prior to the first dose of study drug.
16. A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms).
17. A history of additional risk factors for TdP (e.g., heart failure, hypokalemia, family history of long QT syndrome).
18. The use of concomitant medications that prolong the QT/QTc interval.
19. Patients with the use of strong CYP3A4 inhibitor or inducer.
20. Other malignancies within 5 years except for noninvasive malignancies such as cervical carcinoma in situ, non-melanomatous carcinoma of the skin, or ductal carcinoma in situ of the breast that has been surgically cured. Cancer patients with incidental histologic findings of prostate cancer (tumour/node/metastasis stage T1a or T1b or prostate-specific antigen <10 ng/mL) who have not received hormonal treatment may be included, pending a discussion with the Study Sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-09-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Determination of Recommended Phase 2 Dose (RP2D) | Safety cohort review will be conducted every 4 weeks from the date of first patient's enrollment to review safety data, until all patients have been enrolled and evaluated for toxicity.
  To identify the number of patients who discontinue study drug due to toxicity for each of the two dosing regimens independently.

SECONDARY OUTCOMES:
Adverse Event (AE) | After initiation of study drug, all AEs and SAEs, regardless of attribution, will be collected until 30 days following the last dose of study drug.
  To identify the incidence, severity, and relationship of AEs (as per Common Terminology Criteria for Adverse Events (CTCAE) v 5.0), serious adverse events (SAEs), dose modifications due to AEs.
Objective Response | After initiation of study drug, through time of clinical response.
  To identify the number of patients with clinical benefit (defined as complete response, partial response, or stable disease) and objective response (defined as complete response or partial response) based on the best overall response from tumor evaluations performed every 2 cycles, according to RECIST v1.1, and Duration of Response.
Patient-Reported Outcomes (PRO) | At screening, Day 1 and Day 8 of cycles 1 and 2 (each cycle is 28 days), every 8 weeks after cycle 2, and at the completion of therapy or withdrawal from study, through one month after treatment.
  To identify the incidence, severity, and relationship of AEs using NCI PRO-CTCAE v1.0 questionnaires to evaluate cutaneous, gastrointestinal, visual/perceptual, cardio/circulatory, sleep/wake, and miscellaneous symptoms (as determined by expected toxicity from CX-5461).

OTHER OUTCOMES:
Characterize the molecular profile of tumors and evaluate the predictive value of mutational signatures. | Collected at screening and at the time of disease progression.
  Tumor biopsies are collected from patients to characterize the molecular profile of tumors and evaluate the predictive value of mutational signatures (including BRCA 1/2, PALB2, and other HRD-associated somatic mutations) in predicting response or resistance to CX-5461.
Correlate the significance of changes in ctDNA levels and plasma DNA methylome profiling to detect the evolution of resistant sub-clones and monitor treatment response | Collected at screening, Day 1 and Day 8 of cycles 1 and 2 (each cycle is 28 days), every 8 weeks after cycle 2, and at the time of study discontinuation.
  Blood samples are collected from patients to explore the significance of dynamic changes in ctDNA levels and plasma DNA methylome profiling to detect the evolution of resistant sub-clones and monitor response to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Huang, MD, Study Director — Senhwa Biosciences
Locations (8):
- United States (6):
  - University of California, Los Angeles, Santa Monica, California
  - H. Lee Moffitt Cancer Center and Research Institute Hospital, Tampa, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Ohio State University-James Cancer Hospital and Solove Research Institute, Columbus, Ohio
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
- Canada (2):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No